CLINICAL TRIAL: NCT05709054
Title: The Effect of Manual Therapy Techniques on the Mobility of the Diaphragm in People With Asthma: Protocol for a Randomized Controlled Trial
Brief Title: The Effect of Manual Therapy Techniques on the Mobility of the Diaphragm in People With Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, DIMITRIOS TSIMOURIS, Principal Investigator, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 90853/04-10-2022
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Diaphragm; Breathing retraining; Physiotherapy; Manual therapy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Diaphragmatic excursion assessment with Ultrasonography (Experimental): The time motion mode (M-mode) may be used to measure the diaphragm excursion in a curvilinear low-frequency transducer placed in the midclavicular line and angled in a cranial direction.
  Interventions: Other: Experimental: Diaphragmatic Manual Therapy Group A; Other: Sham Breathing Retraining Exercises Group B
- Chest wall expansion (Experimental): The difference between the values obtained during deep inspiration and expiration will be determined by tape ruler (cm), high degrees represent better outcome, low degrees represent worse outcome.
  Interventions: Other: Experimental: Diaphragmatic Manual Therapy Group A; Other: Sham Breathing Retraining Exercises Group B
- Nijmegen Questionnaire (Experimental): Screening tool used to detect patients with hyperventilation complaints and DB patterns. Scores>20 are used as the cut-score to identify DB in patients with various conditions. NQ values in healthy individuals range from 10 to 12 ± 7 and values do tend to decrease towards these levels after breathing retraining.
  Interventions: Other: Experimental: Diaphragmatic Manual Therapy Group A; Other: Sham Breathing Retraining Exercises Group B
- Asthma Control Test (Experimental): The ACT evaluates how well asthma affects daily functioning, and overall asthma control self-assessment. The score ranges from 5 (poor control of asthma) to 25 (well control of asthma). An ACT score >19 indicates well-controlled asthma.
  Interventions: Other: Experimental: Diaphragmatic Manual Therapy Group A; Other: Sham Breathing Retraining Exercises Group B
- Sf-12v2 questionnaire (Experimental): With one or two questions per domain, it evaluates the exact eight health dimensions as the SF-36v2: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Higher ratings indicate better physical and mental well-functioning, ranging from 0 to 100. It has been suggested that a cut-off of 50 or less be used to identify a physical condition, while a score of 42 or less may signify clinical depression
  Interventions: Other: Experimental: Diaphragmatic Manual Therapy Group A; Other: Sham Breathing Retraining Exercises Group B
- Borg scale (Experimental): The Borg dyspnea scale is a simple, scoring system extensively used to evaluate symptoms of shortness of breath and provides valuable data. It begins with 0, where you have no breathing problems, and rises to 10, where you have the most respiratory distress. As a result, healthcare professionals need to give patients enough time to learn and make sure they comprehend before using it
  Interventions: Other: Experimental: Diaphragmatic Manual Therapy Group A; Other: Sham Breathing Retraining Exercises Group B

INTERVENTIONS:
Other: Experimental: Diaphragmatic Manual Therapy Group A — Experimental: Diaphragmatic Manual Therapy plus Breathing Retraining Exercises group:
  Diaphragm manual therapy will be carried out and consists of a technique intended to stretch and mobilise the diaphragmatic muscle fibers indirectly. The maneuver will be performed in two sets of 10 repetitions, within a 1-minute interval for 10 minutes.
  Breathing retraining exercises will be implemented for 30 minutes, consisting of:
  i) recognition of the abnormal breathing pattern ii) diaphragmatic breathing ii) nose breathing iii) slow breathing and controlled breath holding after exhalation iv) adaptation of the new breathing pattern in everyday life activities and various positions (supine, semi-sitting, sitting) v) breathing control in speech.
Other: Sham Breathing Retraining Exercises Group B — Sham Breathing Retraining Exercises Group B:
  Breathing retraining exercises will be implemented for 30 minutes, consisting of :
  i) recognition of the abnormal breathing pattern ii) diaphragmatic breathing ii) nose breathing iii) slow breathing and controlled breath holding after exhalation iv) adaptation of the new breathing pattern in everyday life activities and various positions (supine, semi-sitting, sitting) v) breathing control in speech.

SUMMARY:
The mechanical alterations related to the overload of respiratory muscles observed in people with persistent asthma can lead to the development of musculoskeletal dysfunctions. Moreover, the produced lung hyperinflation and high lung volumes in the asthma crisis put the diaphragm at a disadvantage in terms of its length-tension curve and lowered its excursion and capacity to generate force. According to a preliminary study, manual therapy (MT) techniques can be used as adjunctive therapy in asthma treatment. The proposed protocol is the first randomized controlled clinical trial to assess MT's efficacy on the diaphragm's ZOA in conjunction with BRE in individuals with well controlled mild moderate and severe asthma. Many musculoskeletal and respiratory outcomes will be used to investigate the under-study therapies' impact.

DETAILED DESCRIPTION:
The diaphragm produces a craniocaudal movement of its dome during contraction, making it the most crucial breathing muscle due to its unique anatomical structure and contribution to minute ventilation (60%-80%). Patients with (COPD) or asthma often develop diaphragmatic dysfunction (DD). This DD is related to the mechanical linkage between its various parts, placing it at a mechanical disadvantage to the muscle fibers. The capacity of the diaphragm to elevate and extend the lower rib cage at the level of the zone of apposition is impaired by this pathological change. This change increases the work of breathing and weakens the diaphragm. People with moderate or severe asthma may experience pulmonary overstretching, which can lead to functional issues. How physiotherapy may increase the mechanical efficiency of the thoracic cage and the effectiveness of the respiratory muscles during breathing has been the main focus of studies in recent decades. Although the use of specific diaphragm MT techniques does not yet have sufficient research documentation, recently published studies reported that there are indications to support their positive effect on pulmonary rehabilitation. The efficacy of diaphragm MT methods has not been investigated in adults with asthma, although it has been investigated in pediatric asthma. The effect of diaphragms MT techniques in combination with BRE has not been investigated. The present study hypothesizes that the combination of the mentioned physiotherapy techniques will contribute positively to the length-tension relationship and mobility of the diaphragm and chest expansion in patients with asthma. Secondary positive improvements are expected in the domain of functionality, (b) the feeling of dyspnea, (c) disease control and (d) abnormal respiratory pattern. The amplification of the above in people with asthma using respiratory standards and applying diaphragm mobilization techniques will contribute to better disease management.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 60 years
* Diagnosed with well controlled asthma (mild, moderate-severe) using spirometry
* No acute exacerbation in the last two months

Exclusion Criteria:

* Cardiopulmonary diseases
* Previous cardiothoracic or abdominal surgery
* Patients who have a recent history of the chest wall or abdominal trauma
* Patients with unstable hemodynamic parameters (arterial pressure >140mmHg systolic and >90mmHg for diastolic inability to understand the verbal commands necessary for the outcome assessments
* Pregnancy
* Neurological diseases
* Previous or parallel participation in interventional programs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic excursion assessment with Ultrasonography | Change from baseline up to 6 weeks and up to 3 months
  The M-mode line is placed at the posterior part of the diaphragm where there is maximal movement and excursion. On the right side, the liver acts as an acoustic window, and the diaphragm is easily identified as a hyperechoic curved line abutting the liver.
Chest wall expansion | Change from baseline up to 6 weeks and up to 3 months
  By placing the tape measure at the level of the axilla (about the level of the sternal angle of Louis), the level of the xiphoid process, or between the xiphoid process and the umbilicus, the therapist identifies the upper, middle, and lower chest wall expansion, respectively. The therapist should repeat the measurement at least three times for each level for higher fidelity.

SECONDARY OUTCOMES:
Nijmegen Questionnaire | Change from baseline up to 6 weeks and up to 3 months
  Screening tool used to detect patients with hyperventilation complaints and DB patterns. Scores>20 are used as the cut-score to identify DB in patients with various conditions. NQ values in healthy individuals range from 10 to 12 ± 7 and values do tend to decrease towards these levels after breathing retraining
Asthma Control Test | Change from baseline up to 6 weeks and up to 3 months
  The ACT evaluates how well asthma affects daily functioning, and overall asthma control self-assessment. The score ranges from 5 (poor control of asthma) to 25 (well control of asthma). An ACT score >19 indicates well-controlled asthma.
Sf-12v2 questionnaire | Change from baseline up to 6 weeks and up to 3 months
  With one or two questions per domain, it evaluates the exact eight health dimensions as the SF-36v2: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Higher ratings indicate better physical and mental well-functioning, ranging from 0 to 100. It has been suggested that a cut-off of 50 or less be used to identify a physical condition, while a score of 42 or less may signify clinical depression
Borg scale | Change from baseline up to 6 weeks and up to 3 months
  The Borg dyspnea scale is a simple, scoring system extensively used to evaluate symptoms of shortness of breath and provides valuable data. It begins with 0, where you have no breathing problems, and rises to 10, where you have the most respiratory distress. As a result, healthcare professionals need to give patients enough time to learn and make sure they comprehend before using it

CONTACTS AND LOCATIONS:
Locations (1):
- Dimitrios Tsimouris, Nea Liosia, Attica, Greece

REFERENCES:
- [Background] Nair A, Alaparthi GK, Krishnan S, Rai S, Anand R, Acharya V, Acharya P. Comparison of Diaphragmatic Stretch Technique and Manual Diaphragm Release Technique on Diaphragmatic Excursion in Chronic Obstructive Pulmonary Disease: A Randomized Crossover Trial. Pulm Med. 2019 Jan 3;2019:6364376. doi: 10.1155/2019/6364376. eCollection 2019. PMID 30719351
- [Background] Rocha T, Souza H, Brandao DC, Rattes C, Ribeiro L, Campos SL, Aliverti A, de Andrade AD. The Manual Diaphragm Release Technique improves diaphragmatic mobility, inspiratory capacity and exercise capacity in people with chronic obstructive pulmonary disease: a randomised trial. J Physiother. 2015 Oct;61(4):182-9. doi: 10.1016/j.jphys.2015.08.009. Epub 2015 Sep 19. PMID 26386894
- [Background] Greising SM, Ottenheijm CAC, O'Halloran KD, Barreiro E. Diaphragm plasticity in aging and disease: therapies for muscle weakness go from strength to strength. J Appl Physiol (1985). 2018 Aug 1;125(2):243-253. doi: 10.1152/japplphysiol.01059.2017. Epub 2018 Apr 19. PMID 29672230
- [Background] Mergoni M, Rossi A. [Physiopathology of acute respiratory failure in COPD and asthma]. Minerva Anestesiol. 2001 Apr;67(4):198-205. Italian. PMID 11376510
- [Background] Santino TA, Chaves GS, Freitas DA, Fregonezi GA, Mendonca KM. Breathing exercises for adults with asthma. Cochrane Database Syst Rev. 2020 Mar 25;3(3):CD001277. doi: 10.1002/14651858.CD001277.pub4. PMID 32212422
- [Background] Grammatopoulou EP, Skordilis EK, Stavrou N, Myrianthefs P, Karteroliotis K, Baltopoulos G, Koutsouki D. The effect of physiotherapy-based breathing retraining on asthma control. J Asthma. 2011 Aug;48(6):593-601. doi: 10.3109/02770903.2011.587583. Epub 2011 Jun 13. PMID 21668321
- [Background] Elnaggar RK, Shendy MA, Mahmoud MZ. Prospective Effects of Manual Diaphragmatic Release and Thoracic Lymphatic Pumping in Childhood Asthma. Respir Care. 2019 Nov;64(11):1422-1432. doi: 10.4187/respcare.06716. Epub 2019 Jul 23. PMID 31337743
- [Background] Vetrugno L, Guadagnin GM, Barbariol F, Langiano N, Zangrillo A, Bove T. Ultrasound Imaging for Diaphragm Dysfunction: A Narrative Literature Review. J Cardiothorac Vasc Anesth. 2019 Sep;33(9):2525-2536. doi: 10.1053/j.jvca.2019.01.003. Epub 2019 Jan 4. PMID 30686657
- [Background] Enrique Leonés-Macías, Irene Torres-Sánchez∗ , Irene Cabrera-Martos, Araceli Ortiz-Rubio, Laura López-López, Marie Carmen Valenza. Effects of manual therapy on the diaphragm in asthmatic patients: A randomized pilot study. International Journal of Osteopathic Medicine; International Journal of Osteopathic Medicine 29 (2018) 26-31DOI: 10.1016/j.ijosm.2018.07.006
- [Derived] Tsimouris D, Grammatopoulou E, Papandreou M, Gioftsos G, Koumantakis G. The effect of manual therapy on diaphragm function in adults with asthma: Protocol for a randomized controlled trial. F1000Res. 2024 Mar 19;12:1361. doi: 10.12688/f1000research.141455.2. eCollection 2023. PMID 39359613
- See also: The Physiotherapy Department of the University of West Attica in Athens, responsible for the coordination of the trial. — http://www.phys.uniwa.gr/
- Available data/document: Clinical Study Report — https://doi.org/10.1016/j.ijosm.2018.07.006